CLINICAL TRIAL: NCT07328139
Title: Comparison of the Effects of Core Stabilization Exercises on Balance and Trunk Endurance in Individuals With Anterior Cruciate Ligament Reconstruction Surgery and Healthy Individuals.
Brief Title: Effects of Core Exercises on Balance in People With and Without ACL Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep HOŞBAY, Head of the Department of Physiotherapy and Rehabilitation, Biruni University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/361
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACL Reconstruction Group (Experimental): Participants in this arm are individuals who have undergone unilateral Anterior Cruciate Ligament (ACL) reconstruction surgery within the last 5 years. These participants will receive a core stabilization exercise program for 8 weeks, with supervised sessions held twice per week. The exercise program includes movements such as the Hundreds, clam exercise, plank, side plank, dead bug, and bridging.
  Interventions: Behavioral: Core Stabilization Exercise Program
- Healthy Control Group (Active Comparator): Participants in this arm are healthy individuals with no known history of lower extremity injury or surgery. This group is matched to the ACL Reconstruction Group. These participants will also receive the same core stabilization exercise program for 8 weeks, with supervised sessions held twice per week, to serve as a comparison group.
  Interventions: Behavioral: Core Stabilization Exercise Program

INTERVENTIONS:
Behavioral: Core Stabilization Exercise Program — Participants receive a supervised core stabilization exercise program for a duration of 8 weeks. Sessions are conducted twice per week by a physiotherapist. The program includes a set of standardized exercises such as the Hundreds, clam exercise, plank, side plank, dead bug exercise, curl-ups, and bridging.

SUMMARY:
The main purpose of this study is to evaluate and compare the effects of an 8-week core stabilization exercise program on balance, trunk muscle endurance, and lower body strength.

The study includes two groups of participants: 15 individuals who have had Anterior Cruciate Ligament (ACL) reconstruction surgery and 15 healthy individuals. Both groups will perform the same core stabilization exercises for 8 weeks, twice a week, under the supervision of a physiotherapist.

The goal is to determine if this exercise program improves balance and core strength in people who have had ACL surgery and to compare these results with those of healthy individuals performing the same exercises.

ELIGIBILITY:
Inclusion Criteria

* Aged between 18 and 65 years.
* Agreement to participate regularly in the 8-week exercise program.
* No contraindications to physical activity, as assessed by a medical professional.
* ACLR group: history of unilateral ACL reconstruction within the past five years.
* Control group: no known history of lower extremity injury or surgery.

Exclusion Criteria

* Any musculoskeletal or neurological condition affecting balance or core stabilization.
* Participation in a structured core stabilization exercise program within the previous six months.
* Any acute injury or systemic disease that may interfere with study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Change in Dynamic Balance as Measured by the Y-Balance Test | Baseline and 8 weeks
  The Y-Balance Test (YBT) is used to assess dynamic postural control. Participants stand on one leg at the center of a grid and reach with the other leg as far as possible in three directions: anterior, posteromedial, and posterolateral. The maximum reach distance in each direction is recorded in centimeters. A higher score indicates better dynamic balance.
Change in Trunk Muscle Endurance as Measured by the McGill Core Endurance Tests | Baseline and 8 weeks
  Trunk muscle endurance is assessed using the McGill Core Endurance Test battery, which consists of four tests: a trunk flexor endurance test, a trunk extensor endurance test (Sorenson test), and right and left lateral trunk muscle endurance tests (side bridge). The time in seconds that a participant can hold each specific position without losing the correct form is recorded. A longer time indicates greater endurance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Faculty of Medicine Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No